CLINICAL TRIAL: NCT06296459
Title: Radiographic Changes in the Maxillary Sinus Following Closed Sinus Augmentation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20220556HU
Record Dates: First submitted 2024-02-28; First posted 2024-03-06 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Dental Implant
Keywords: Cone beam computed tomography; Sinus anatomy; Dental implant placement

STUDY DESIGN:
Intervention Model Description: A 2 arm study using two methods of imaging in a participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low volume CBCT (Active Comparator): Radiographic low volume cone beam computed tomography used to plan implant placement
  Interventions: Other: 3D R100 scanner
- Standard periapical radiographs (Placebo Comparator): Standard radiography used to plan implant placement
  Interventions: Other: Conventional Radiograph

INTERVENTIONS:
Other: 3D R100 scanner — A cone beam computed tomography used for planning of implant surgery
  Other Names: Veraviewpocs
  Arms: Low volume CBCT
Other: Conventional Radiograph — Imaging used as standard of care to plan for implant surgery
  Other Names: Standard Periapical Radiograph
  Arms: Standard periapical radiographs

SUMMARY:
A closed sinus augmentation is performed for dental implant placement.

DETAILED DESCRIPTION:
Patients who are diagnosed as needing sinus augmentation by a closed approach for dental implant placement will be recruited. A cone beam computed tomography (CBCT) study is the standard of care prior to dental implant placement. However, following closed sinus augmentation nothing is known as to the extent of augmentation in the medial to lateral (cross-sectional) dimension. Patients will have a low volume CBCT taken immediately postsurgically, and again at the six-month postoperative visit to determine the dimensional changes in the augmentation. These images will be compared to standard periapical radiographs at the same time points.

ELIGIBILITY:
Inclusion Criteria:

1. Partially edentulous patients (18-85 years of age) requiring maxillary sinus augmentation for dental implant placement.
2. At least 5mm of native bone below the maxillary sinus.
3. Nonsmokers.
4. If diabetic, current HbA1C <7.0 (less than or equal to 7.0)

Exclusion Criteria:

1. Maxillary sinus disease.
2. Pregnancy or attempting to become pregnant.
3. Diseases that affect bone metabolism.
4. Use of medications known to affect bone metabolism.
5. Tobacco use.
6. Alcoholism or recreational drug use.
7. Diabetic with HbA1C >7.0 (above 7.0)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-09-21 (Actual); Primary Completion 2024-12-19 (Actual); Study Completion 2024-12-19 (Actual)

PRIMARY OUTCOMES:
Dimensional Change in augmentation at 8mm | Baseline immediately postoperatively and at 6 months
  Determine the morphologic changes to maxillary sinus anatomy three dimensionally when a closed sinus augmentation is performed for dental implant placement at 8mm from alveolar crest.
Dimensional Change in augmentation at 10mm | Baseline immediately postoperatively and at 6 months
  Determine the morphologic changes to maxillary sinus anatomy three dimensionally when a closed sinus augmentation is performed for dental implant placement at 10 mm from alveolar crest.
Dimensional Change in augmentation at 12mm | Baseline immediately postoperatively and at 6 months
  Determine the morphologic changes to maxillary sinus anatomy three dimensionally when a closed sinus augmentation is performed for dental implant placement at 12 mm from alveolar crest.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Powell, DDS, MS, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- The University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
All deidentified participant data will be shared with colleagues
Supporting Information: Study Protocol, SAP
Time Frame: After study completion in a peer review journal